CLINICAL TRIAL: NCT06680076
Title: Observational Study of Changes in Plasma and Intestinal Mucosa Lipid Profiles in Patients With Inflammatory Bowel Disease
Brief Title: Study on Lipid Profile Changes in Plasma and Intestinal Mucosa of Patients With Inflammatory Bowel Disease
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Hongyu Xu, Chief of the GI department, First Affiliated Hospital of Harbin Medical University
Other Study IDs: Harbin Medical University
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD; lipid metabolism; activity
MeSH Terms: conditions — Inflammatory Bowel Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colon tissue and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease group: Patients who have inflammation bowel disease.
- Health group: Healthy people who volunteered to participate.

SUMMARY:
This study aimed to demonstrate the characteristic lipid profile changes in patients with inflammatory bowel disease.

DETAILED DESCRIPTION:
This study aimed to demonstrate the characteristic lipid profile changes in patients with inflammatory bowel disease.

The investigators followed up with patients with different stages of IBD and collected plasma and lesion tissues from patients and healthy volunteers for lipid metabolism-related substances to assess the changes in lipid metabolism in patients with different stages of IBD and their impact on disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease; aged 18-80 years; all cases agreed to participate in the study.
* Healthy volunteers who agreed to participate in the study.

Exclusion Criteria:

* Patients with severe heart disease; patients with severe kidney disease; patients with low blood pressure; patients with severe infections such as sepsis or pneumonia; patients who have used immunosuppressants such as 6-mercaptopurine, imidazole thiopurine, and cyclosporine within a short period, and women during pregnancy; patients who are post-colon resected; patients who disagreed to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients who have inflammation bowel disease.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Differential lipid composition between disease and healthy groups | 14 weeks
  Differences in lipid composition between disease and healthy groups.
Differences in lipid composition between active and remission disease | 14 weeks
  Differences in lipid composition between active and remission disease

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu D Xu, PHD, Study Director — Harbin Medical University
Locations (1):
- Carol, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No